CLINICAL TRIAL: NCT02378857
Title: Fontan Circulation and Cardiopulmonary Function: Prognostic Factors, Hemodynamics and Long-term Effects
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Thomas Möller, Senior consultant pediatric cardiologist, MD PhD, Oslo University Hospital
Other Study IDs: 2013/1331 (REK); 2014077 (Other: South-Eastern Norway Regional Health Authority)
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Congenital Heart Disease
Keywords: Univentricular heart defect; Fontan circulation
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — EDTA, citrate and serum samples for analysis for vitamin status, biochemical analysis, inflammation markers and organ specific markers.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patient group: Adolescents (15-18 years of age) With univentricular heart defects and Fontan type palliation.
- Control group: Age- and gender-matched healthy individuals

SUMMARY:
Cross-sectional study of a national cohort of adolescents with univentricular congenital heart defects and Fontan type palliation.

DETAILED DESCRIPTION:
A study group of 40-50 individuals will be investigated by non-invasive and invasive methods, including echocardiography at rest and during exercise, heart catheterization with advanced hemodynamic studies, cardiac and abdominal MRI, abdominal ultrasound and transient elastography, quality of life assessment and cardiopulmonary exercise testing. A selection of tests will be performed in a healthy control group as well.

ELIGIBILITY:
Inclusion Criteria:

* age, heart defect, heart surgery and type of palliation/correction, informed consent

Exclusion Criteria:

* non-consenting, contraindications or increased risk to perform study tests (i.e. metal parts prohibiting MRI, motoric impairment prohibiting CPET)

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All adolescents i Norway with univentricular heart defects and Fontan type palliation
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-03; Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Hemodynamic status | Current at time of inclusion
  Status as found by invasive and non-invasive assessment
Structural and functional hepatic changes | Current at time of inclusion
  Status as found by non-invasive assessment
Cardio-pulmonary function and functional reserve | Current at time of inclusion
  Status as found by non-invasive assessment
Quality of life and psycho-social outcome | Current at time of inclusion
  Status as found by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Moller, MD PhD, Principal Investigator — Oslo University Hospital, University of Oslo
Locations (1):
- Oslo University Hospital, Rikshospitalet, Department of Paediatric Cardiology, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moller T, Klungerbo V, Diab S, Holmstrom H, Edvardsen E, Grindheim G, Brun H, Thaulow E, Kohn-Luque A, Rosner A, Dohlen G. Circulatory Response to Rapid Volume Expansion and Cardiorespiratory Fitness in Fontan Circulation. Pediatr Cardiol. 2022 Apr;43(4):903-913. doi: 10.1007/s00246-021-02802-y. Epub 2021 Dec 17. PMID 34921324